CLINICAL TRIAL: NCT00424203
Title: Multicenter Pilot Clinical Study of Adjuvant Chemotherapy for Subjects Over 70 Years: Impact on the Independence and Quality of Life of the Administration of Anthracycline-Based Chemotherapy in Adjuvant Setting for Patients Presenting With Immediately Operable Breast Cancer, Hormone Receptor Negative (RH-), and Lymph Node Positive (pN+) or pN0 But of Scarff-Bloom-Richardson* Grade III and ≥ 2cm [GERICO]
Brief Title: Doxorubicin and Cyclophosphamide in Treating Older Women With Stage I, Stage II, or Stage III Breast Cancer That Has Been Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000523419; FRE-FNCLCC-GERICO-06-0502; EU-20667; EUDRACT-2005-000069-20
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Breast Cancer; Cognitive/Functional Effects; Depression; Malnutrition; Psychosocial Effects of Cancer and Its Treatment
Keywords: cognitive/functional effects; depression; malnutrition; psychosocial effects of cancer and its treatment; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; estrogen receptor-negative breast cancer; progesterone receptor-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Depression; Malnutrition | interventions — Cyclophosphamide; Doxorubicin; Chemotherapy, Adjuvant; Mental Status and Dementia Tests; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Myocet, Endoxan (Experimental)
  Interventions: Drug: AC regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Procedure: adjuvant therapy; Procedure: cognitive assessment; Procedure: management of therapy complications; Procedure: psychosocial assessment and care; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: AC regimen
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Procedure: adjuvant therapy
Procedure: cognitive assessment
Procedure: management of therapy complications
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving combination chemotherapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving doxorubicin together with cyclophosphamide works in treating older women with stage I , stage II, or stage III breast cancer that has been removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the independence of older women with resected stage I, II, or III breast cancer treated with adjuvant doxorubicin hydrochloride and cyclophosphamide.

Secondary

* Determine the impact of this regimen on other aspects of the patient's life, utilizing the Comprehensive Geriatric Assessment, the Mini-Nutritional Assessment, the Folstein Mini-Mental State Exam, the Geriatric Depression Scale, and the Cumulative Illness Rating Scale-Geriatrics.
* Determine the quality of life of patients treated with this regimen.
* Determine the acceptability of this regimen in these patients.
* Determine the toxicity of this regimen, in terms of cardiac issues and anemia, in these patients.
* Determine recurrence-free survival, event-free survival, and overall survival of patients treated with this regimen.

OUTLINE: This is a pilot, nonrandomized, multicenter study.

Patients receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients complete questionnaires at baseline and after completion of chemotherapy. Questionnaires include the Comprehensive Geriatric Assessment, the Mini-Nutritional Assessment (malnutrition), the Folstein Mini-Mental State Exam (cognitive function), the Geriatric Depression Scale (depression), the Cumulative Illness Rating Scale - Geriatrics (comorbidities), and the EORTC Quality of Life Questionnaire Core 30 (quality of life).

After completion of study therapy, patients are followed every 3 months for 4 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive adenocarcinoma of the breast

  * Stage I, II or III disease

    * pN+ or pN0 with grade III disease (tumor size ≥ 2 cm)
    * No metastatic disease
* Must have undergone prior conservative or radical surgery that included axillary lymph node or sentinel node dissection

  * No residual tumor
  * Negative margins
* Hormone receptor status:

  * Estrogen receptor and progesterone receptor negative

PATIENT CHARACTERISTICS:

* Female
* Postmenopausal
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 100,000/mm³
* Hemoglobin > 10 g/dL
* Alkaline phosphatase < 2.5 times upper limit of normal (ULN)
* Bilirubin < 1.25 times ULN
* AST and ALT < 2.5 times ULN
* Creatinine clearance ≥ 40 mL/min
* No contraindication to receiving anthracyclines or alkalizing agents
* FEV normal
* Activities of Daily Living (ADL) score ≥ 5

  * No decrease of ≥ 1 point within the past 3 months
* None of the following at baseline:

  * Cognitive deficiency (Folstein Mini-Mental State < 25)
  * Severe depression (Geriatric Depression Scale ≥ 20)
  * Severe malnutrition (Mini-Nutritional Assessment ≤ 17)
* No other serious comorbid condition (Cumulative Illness Rating Scale - Geriatrics grade 3-4), including any of the following:

  * Cardiac insufficiency
  * Unstable angina
  * Myocardiopathy
  * Myocardial infarction within the past year
  * Uncontrolled hypertension
  * Uncontrolled high-risk arrhythmia
  * Severe medullary insufficiency
  * Neurological or psychological condition that would preclude study consent
  * Uncontrolled or active infection
  * Severe urinary tract infection
  * Preexisting hematuria
  * Active ulcer
  * Uncontrolled diabetes
* No other cancer within the past 5 years except for basal cell skin cancer or carcinoma in situ of the cervix
* No familial, geographical, social, or psychological condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 60 days since prior therapeutic surgery
* At least 4 weeks since prior investigational drugs

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients maintaining their independence as assessed by Activities of Daily Living (ADL) score on 6 items after the fourth course of chemotherapy | 12 weeks

SECONDARY OUTCOMES:
Impact of adjuvant chemotherapy on ADL score, quality of life, treatment acceptability, toxicity, and survival (recurrence-free, progression-free, and overall survival) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: E. G. C. Brain, MD, PhD, Study Chair — Institut Curie
Locations (17):
- France (17):
  - Centre Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Institut Bergonie, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Hopital Perpetuel Secours, Levallois-Perret
  - Centre Leon Berard, Lyon
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
  - Hopital Europeen Georges Pompidou, Paris
  - Institut Curie Hopital, Paris
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Rene Huguenin, Saint-Cloud
  - C.H. Senlis, Senlis
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy